CLINICAL TRIAL: NCT05488197
Title: The Value of Second-trimester Uterine Artery Doppler Analysis in the Prediction of GDM in a Low- Risk Population
Acronym: PS-GDM-2022
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Filiz Yarsilikal Guleroglu, Medical Doctor, Haseki Training and Research Hospital
Other Study IDs: PS-GDM-2022; PS-GDM-2022 (Other)
Record Dates: First submitted 2022-07-28; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 participants with gestational diabetes
  Interventions: Other: uterine artery doppler at 18-23 weeks of pregnancy
- Group 2 participants without gestational diabetes
  Interventions: Other: uterine artery doppler at 18-23 weeks of pregnancy

INTERVENTIONS:
Other: uterine artery doppler at 18-23 weeks of pregnancy — uterine artery doppler at 18-23 weeks of pregnancy

SUMMARY:
In the current literature, there are not enough studies related to the use of uterine artery Doppler indices in the second trimester for the prediction of GDM. Considering that it may be useful in the prediction of GDM in low-risk patient groups for GDM, it was found useful to consider uterine artery Doppler analysis within the scope of this study.In this study, the investigators aimed to assess the value of second-trimester uterine artery Doppler analysis in the prediction of GDM in a low- risk population.

DETAILED DESCRIPTION:
This retrospective research was conducted between June 2020 and December 2021 at the Perinatology Clinic of Haseki Training and Research Hospital. Maternal age between 18 and 42 years and gestational age between 18 and 23 weeks were the inclusion criteria.Pregnant women's computerized records were used to compare the relevant data of women diagnosed with gestational diabetes and women with normal glucose tolerance . Transabdominal ultrasonography was performed for anatomical scanning, and the uterine artery Doppler was obtained using ultrasonographic devices with a 2.0-7.0 megahertz convex probe. The uterine artery waveforms were obtained using pulsed-wave Doppler with an insonation angle of 30° and a peak systolic velocity greater than 60 cm/s. Three identical waveforms were obtained consecutively on each side. In addition to recording the presence or absence of notching, the mean uterine artery pulsatility index (UAPI) was also obtained. Abnormal uterine artery Doppler was defined as a mean UAPI greater than the 95th percentile for each gestation.Increased uterine artery pulsatility index and/or diastolic notch in the uterine artery between 18-23 weeks of pregnancy can predict the risk of GDM in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant women with or without Gestational Diabetes in low- risk population

Exclusion Criteria:

* Pregestational Diabetes
* Preeclampsia
* Intrauterine growth restriction
* Chronic Maternal Disease

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women with or without Gestational Dibetes in low- risk population
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Uterine artery Doppler ultrasonography in gestational diabetes mellitus | Through study completion, an average of 18 months
  To investigate and compare uterine artery pulsatility index by Doppler ultrasonography in patients with gestational diabetes mellitus (GDM) and without to non-diabetic controls.

SECONDARY OUTCOMES:
Prediction of GDM with uterine artery pulsatility index cut-offs | Through study completion, an average of 18 months
  Cut off values of uterine artery pulsatility index will be estimated to predict GDM

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)